CLINICAL TRIAL: NCT05586113
Title: The Efficacy of Bismuth-containing Quadruple Therapy in the First-line Treatment of Helicobacter Pylori Infection in 10 Days and 14 Days: a Prospective, Randomized, Controlled Study
Brief Title: The Efficacy of 10-day or 14-day Course of Bismuth-containing Quadruple Therapy:A Randomized Clinical Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong University (Other)
Collaborators: Linyi People's Hospital (Other); Weifang Medical University (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, Director of Qilu Hospital gastroenterology department, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-SDU-QILU-G005
Record Dates: First submitted 2022-10-17; First posted 2022-10-19 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Helicobacter Pylori Infection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10-day treatment group (Experimental): 10-day Tegoprazan bismuth-containing quadruple therapy Tegoprazan（Luo Xin Pharmaceutical Group Co. LTD）50mg bid Amoxicillin (Amoxicillin, United Laboratories Co., LTD) 1000mg bid Tetracycline (Huanan Brand, Guangdong Huanan Pharmaceutical Co. LTD.) 500mg qid Bismuth potassium Citrate (Lizhu Delle, Lizhu Group Pharmaceutical Factory) 2g bid
  Interventions: Drug: 10-day Tegoprazan bismuth-containing quadruple therapy
- 14-day treatment group (Active Comparator): 14-day Tegoprazan bismuth-containing quadruple therapy Tegoprazan（Luo Xin Pharmaceutical Group Co. LTD）50mg bid Amoxicillin (Amoxicillin, United Laboratories Co., LTD) 1000mg bid Tetracycline (Huanan Brand, Guangdong Huanan Pharmaceutical Co. LTD.) 500mg qid Bismuth potassium Citrate (Lizhu Delle, Lizhu Group Pharmaceutical Factory) 2g bid
  Interventions: Drug: 10-day Tegoprazan bismuth-containing quadruple therapy

INTERVENTIONS:
Drug: 10-day Tegoprazan bismuth-containing quadruple therapy — 10-day Tegoprazan bismuth-containing quadruple therapy: Tegoprazan（Luo Xin Pharmaceutical Group Co. LTD）50mg bid Amoxicillin (Amoxicillin, United Laboratories Co., LTD) 1000mg bid Tetracycline (Huanan Brand, Guangdong Huanan Pharmaceutical Co. LTD.) 500mg qid Bismuth potassium Citrate (Lizhu Delle, Lizhu Group Pharmaceutical Factory) 2g bid

SUMMARY:
The researchers collect treatment-naive H.pylori-positive patients from the outpatient clinic. The subjects were randomized to receive a 10-day or 14-day course of Tegoprazan bismuth-containing quadruple eradication therapy at 6 weeks after treatment, subjects underwent another 13C-urea breath test. Calculate the eradication rates, adverse reaction rates, patient compliance and cost-effectiveness index of each group.

DETAILED DESCRIPTION:
The researchers collect treatment-naive H.pylori-positive patients from the outpatient clinic. If the subject meets the selection criteria but not the exclusion criteria, and signs an informed consent form, the researchers randomized the subjects in groups: subjects received a 10-day or 14-day course of Tegoprazan bismuth-containing quadruple eradication therapy. The medication of groups are as follows. 6-8 weeks after the eradication treatment, the subjects will review the 13C-urea breath test, and the researcher records the results.

After all subjects were tested, the eradication rates, adverse reaction rates, patient compliance and cost-effectiveness index of each group were calculated.

According to the course of treatment, it is randomized into a 10-day treatment group and a 14-day treatment group. The two groups of bismuth quadruple regimens are the same, as follows:

Amoxicillin 1000mg bid+ Tetracycline 500mg qid+ Bismuth + Tegoprazan 50mg bid

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-70.
* Patients with H.pylori infection (Positive for any of the following: 13C/14C-urea breath test, histopathology test, rapid urease test, stool H.pylori antigen test).
* Patients who have not previously received helicobacter pylori eradication therapy

Exclusion Criteria:

* Patients with serious underlying diseases, such as liver insufficiency (Aspartate aminotransferase or alanine aminotransferase greater than 1.5 times the normal value), renal insufficiency (Cr≥2.0mg/dL or glomerular filtration rate <50 ml/min), immunosuppression, malignant tumors, Coronary heart disease or coronary artery stenosis ≥75%.
* Patients who are pregnant or lactating or unwilling to take contraceptive measures during the trial.
* Patients with active gastrointestinal bleeding.
* Patients with a history of upper gastrointestinal surgery.
* Patients allergic to treatment drugs.
* Patients with medication history of bismuth agents, antibiotics, proton pump inhibitor and other drugs within 4 weeks
* Patients with other behaviors that may increase the risk of illness, such as alcohol and drug abuse
* Patients who are unwilling or incapable to provide informed consents.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 398 (Estimated)
Dates: Start 2023-02-06 (Estimated); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Eradication rate | immediately after the procedure
  Both intention to treat (ITT) and per-protocol (PP) analyses will be used for the assessment of the eradication rates of Helicobacter pylori infections in two groups. The ITT analysis includes all randomly assigned patients who take at least one dose of the study medications. The PP analysis is limited to patients who take over 90% of the study medications and complete follow-up.

SECONDARY OUTCOMES:
Rate of adverse reactions | immediately after the procedure
  Rate of adverse reactions
Patient compliance | immediately after the procedure
  Good compliance is defined as the actual dosage is within the range of 80%-100% of the dosage that should be taken.
Cost-effectiveness index | immediately after the procedure
  Ratio of costs to effectiveness

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu hosipital, Jinan, Shandong, China

REFERENCES:
- [Background] Du LJ, Chen BR, Kim JJ, Kim S, Shen JH, Dai N. Helicobacter pylori eradication therapy for functional dyspepsia: Systematic review and meta-analysis. World J Gastroenterol. 2016 Mar 28;22(12):3486-95. doi: 10.3748/wjg.v22.i12.3486. PMID 27022230
- [Background] Alba C, Blanco A, Alarcon T. Antibiotic resistance in Helicobacter pylori. Curr Opin Infect Dis. 2017 Oct;30(5):489-497. doi: 10.1097/QCO.0000000000000396. PMID 28704226
- [Background] Hooi JKY, Lai WY, Ng WK, Suen MMY, Underwood FE, Tanyingoh D, Malfertheiner P, Graham DY, Wong VWS, Wu JCY, Chan FKL, Sung JJY, Kaplan GG, Ng SC. Global Prevalence of Helicobacter pylori Infection: Systematic Review and Meta-Analysis. Gastroenterology. 2017 Aug;153(2):420-429. doi: 10.1053/j.gastro.2017.04.022. Epub 2017 Apr 27. PMID 28456631
- [Background] Liu WZ, Xie Y, Lu H, Cheng H, Zeng ZR, Zhou LY, Chen Y, Wang JB, Du YQ, Lu NH; Chinese Society of Gastroenterology, Chinese Study Group on Helicobacter pylori and Peptic Ulcer. Fifth Chinese National Consensus Report on the management of Helicobacter pylori infection. Helicobacter. 2018 Apr;23(2):e12475. doi: 10.1111/hel.12475. Epub 2018 Mar 7. PMID 29512258
- [Background] Malfertheiner P, Megraud F, O'Morain CA, Gisbert JP, Kuipers EJ, Axon AT, Bazzoli F, Gasbarrini A, Atherton J, Graham DY, Hunt R, Moayyedi P, Rokkas T, Rugge M, Selgrad M, Suerbaum S, Sugano K, El-Omar EM; European Helicobacter and Microbiota Study Group and Consensus panel. Management of Helicobacter pylori infection-the Maastricht V/Florence Consensus Report. Gut. 2017 Jan;66(1):6-30. doi: 10.1136/gutjnl-2016-312288. Epub 2016 Oct 5. PMID 27707777
- [Background] Liou JM, Malfertheiner P, Lee YC, Sheu BS, Sugano K, Cheng HC, Yeoh KG, Hsu PI, Goh KL, Mahachai V, Gotoda T, Chang WL, Chen MJ, Chiang TH, Chen CC, Wu CY, Leow AH, Wu JY, Wu DC, Hong TC, Lu H, Yamaoka Y, Megraud F, Chan FKL, Sung JJ, Lin JT, Graham DY, Wu MS, El-Omar EM; Asian Pacific Alliance on Helicobacter and Microbiota (APAHAM). Screening and eradication of Helicobacter pylori for gastric cancer prevention: the Taipei global consensus. Gut. 2020 Dec;69(12):2093-2112. doi: 10.1136/gutjnl-2020-322368. Epub 2020 Oct 1. PMID 33004546
- [Background] Dore MP, Farina V, Cuccu M, Mameli L, Massarelli G, Graham DY. Twice-a-day bismuth-containing quadruple therapy for Helicobacter pylori eradication: a randomized trial of 10 and 14 days. Helicobacter. 2011 Aug;16(4):295-300. doi: 10.1111/j.1523-5378.2011.00857.x. PMID 21762269
- [Background] Cho YK, Choi MG, Choi SC, Lee KM, Kim TO, Park SH, Moon JS, Lim YJ, Kang DH, Cheon GJ, Baik GH, Kim KO, Cho KB, Jang JS, Park JJ, Son BK, Jung HK, Kim BW, Kim SK, Lee ST, Cha JM, Kim AR, Kim EJ, Park HW, Song GS. Randomised clinical trial: tegoprazan, a novel potassium-competitive acid blocker, or lansoprazole in the treatment of gastric ulcer. Aliment Pharmacol Ther. 2020 Sep;52(5):789-797. doi: 10.1111/apt.15865. Epub 2020 Jul 23. PMID 32701188
- [Background] Choi YJ, Lee YC, Kim JM, Kim JI, Moon JS, Lim YJ, Baik GH, Son BK, Lee HL, Kim KO, Kim N, Ko KH, Jung HK, Shim KN, Chun HJ, Kim BW, Lee H, Kim JH, Chung H, Kim SG, Jang JY. Triple Therapy-Based on Tegoprazan, a New Potassium-Competitive Acid Blocker, for First-Line Treatment of Helicobacter pylori Infection: A Randomized, Double-Blind, Phase III, Clinical Trial. Gut Liver. 2022 Jul 15;16(4):535-546. doi: 10.5009/gnl220055. Epub 2022 Jul 6. PMID 35791797
- [Background] Kim SY, Lee SW, Jung SW, Koo JS, Yim HJ, Park JJ, Chun HJ, Lee HS, Choi JH, Kim CD, Ryu HS. Comparative study of Helicobacter pylori eradication rates of twice-versus four-times-daily amoxicillin administered with proton pump inhibitor and clarithromycin: a randomized study. Helicobacter. 2008 Aug;13(4):282-7. doi: 10.1111/j.1523-5378.2008.00615.x. PMID 18665938